CLINICAL TRIAL: NCT01259856
Title: Randomized Trial of Pegylated Interferon Alfa-2a Versus Hydroxyurea Therapy in the Treatment of High Risk Polycythemia Vera (PV) and High Risk Essential Thrombocythemia (ET)
Brief Title: Randomized Trial of Pegylated Interferon Alfa-2a Versus Hydroxyurea in Polycythemia Vera (PV) and Essential Thrombocythemia (ET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ronald Hoffman (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH); Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Ronald Hoffman, Professor of Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 09-1300-00002; P01CA108671 (NIH); MPD-RC 112 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2010-12-07; First posted 2010-12-14 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: High Risk Polycythemia Vera; High Risk Essential Thrombocythemia
Keywords: Polycythemia vera; Essential thrombocythemia; Hydroxyurea; PEGASYS; Pegylated Interferon Alfa-2a
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential | interventions — peginterferon alfa-2a; Hydroxyurea; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEGASYS (Experimental): The subject will begin receiving the PEGASYS at a dose level of 45 micrograms weekly and gradually get increased to the maximum dose of 180 micrograms per week. The dose will be administered by prefilled syringes that will be injected subcutaneously. Subjects will receive therapy for up to 12 months.
  Interventions: Drug: PEGASYS; Drug: Aspirin
- Hydroxyurea (Active Comparator): Subjects will receive a 500mg tablet to be taken twice daily for up to 12 months of treatment.
  Interventions: Drug: Hydroxyurea; Drug: Aspirin

INTERVENTIONS:
Drug: PEGASYS — The subject will begin receiving the PEGASYS at a dose level of 45 micrograms weekly and gradually get increased to the maximum dose of 180 micrograms per week. The dose will be administered by prefilled syringes that will be injected subcutaneously. Subjects will receive therapy for up to 12 months.
  Other Names: Pegylated Interferon Alfa-2a
  Arms: PEGASYS
Drug: Hydroxyurea — Subjects will receive a 500mg tablet to be taken twice daily for up to 12 months of treatment.
  Other Names: Hydroxycarbamide
  Arms: Hydroxyurea
Drug: Aspirin — Subject will be asked to take 81 to 100mg per day for the 12 months of the study treatment.
  Other Names: acetylsalicylic acid

SUMMARY:
This research is looking at two conditions, Essential Thrombocythemia (ET) and Polycythemia Vera (PV). ET causes people to produce too many blood cells called platelets and PV causes too many platelets and red blood cells to be made. Platelets are particles which circulate in the blood stream and normally prevent bleeding and bruising. Having too many platelets in the blood increases the risk of developing blood clots, which can result in life threatening events like heart attacks and strokes. When the number of red blood cells is increased in PV this will slow the speed of blood flow in the body and increases the risk of developing blood clots.

The purpose of this study is to look at the effectiveness of giving participants who have been diagnosed with ET or PV one of two different study regimens over time. The study subject will be followed for their condition for about 5 years. The subject will be randomized into one of two study regimens, either Pegylated Interferon Alfa-2a (PEGASYS) or Aspirin and Hydroxyurea (also called Hydroxycarbamide). The subject must be newly diagnosed or already receiving treatment for either PV or ET. Each of the study drugs used in this study is already being used to treat subjects with ET or PV currently, but the investigators are unsure which study drug is better.

DETAILED DESCRIPTION:
The Philadelphia chromosome negative myeloproliferative neoplasms (MPN) are a group of clonal hematological malignancies that are characterized by a chronic course which can be punctuated by a number of disease related events including thrombosis, hemorrhage, pruritis and leukemic transformation. These disorders include Polycythemia Vera (PV), Essential Thrombocythemia (ET) and Primary Myelofibrosis (PM). Recently an acquired somatic mutation in the intracellular kinase, JAK2 (JAK2V617F) has been observed in 95% of patients with PV, 50% of patients with ET and 50% of patients with primary myelofibrosis. At present the chemotherapeutic agent hydroxyurea is the standard of care for high risk patients with PV. Concern exists about prolonged use of this drug leading to leukemia and the inability of hydroxyurea to eliminate the malignant clone.

Interferon (rIFN -2b), is a drug that appears to be non-leukemogenic, and may have a preferential activity on the malignant clone in PV, as suggested by cytogenetic remissions obtained in patients treated with rIFN -2b. Several investigators recently reported that patients with PV treated with rIFN -2b had lower JAK2V617F allele burdens as compared to a control group that included patients treated with phlebotomy, hydroxyurea, or anagrelide, or who remained untreated. The results confirm the hypothesis that rIFN -2b preferentially targets the malignant clone in PV and raises the possibility that the JAK2V617F allele burden, and a reversion of clonal hematopoiesis monitored in females by expression of X-chromosome polymorphic alleles maybe useful in monitoring minimal residual disease in PV patients.

Pegylated Interferon Alfa-2a (PEGASYS) has been demonstrated in phase II trials of patients with PV and ET to have clinical efficacy as measured by normalization of myeloproliferation, lack of vascular events while on therapy, and a decrease in the JAK2V617F allele burden. Overall the tolerability of the therapy was good, with each of these trials having a dropout rate secondary to toxicity of less than 10% of those enrolled. Although dropout rates for toxicity were low, that is not to say the therapy was without symptomatic toxicity, and indeed a spectrum of toxicities might be encountered and need to be weighed in the analysis of the net clinical benefit patients experience on a clinical trial with Pegylated Interferon Alfa-2a.

A new MPN assessment form will be utilized in this study. This 19 item instrument includes a previously validated 9 item brief fatigue inventory (BFI), symptoms related to splenomegaly, inactivity, cough, night sweats, pruritus, bone pains, fevers, weight loss, and an overall quality of life assessment. The instrument yields an independent result for each symptom (fatigue is a composite score), as this methodology (of linear analog scale assessment [LASA]) has proven very valid in the past. This instrument was validated prospectively (by comparison to a panel of instruments each containing an aspect of the MPN-SAF) for administration at a single time point.

This is a randomized trial between hydroxyurea and Pegylated Interferon Alfa-2a, it is an open label clinical trial in two independent disease strata: (1) high risk polycythemia vera and (2) high risk essential thrombocythemia.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Essential Thrombocythemia (ET) or Polycythemia Vera (PV) shall be made in accordance with the WHO (2008)criteria (Swerdlow 2008) as shown below.
* Diagnosis < 5 years prior to entry.
* Polycythemia Vera (2 major criteria required)

  1. Hb >18.5g/dl (♂) or 16.5g/dl (♀) or HCT >99 percentile reference range or Elevated red cell mass (>25% above mean predicted value) or Hb >17g/dl (♂) or 15g/dl (♀) if associated with a sustained rise from baseline with no apparent cause (e.g. treated iron deficiency).
  2. Presence of JAK2V617F

     * If source documentation of diagnostic criterion #1 cannot be obtained, then diagnosis can be made with (1) the addition of an erythropoietin level below the reference range of normal AND (2) bone marrow biopsy showing hypercellularity for age with trilineage (panmyelosis) with prominent erythroid, granulocytic, and megakaryocytic proliferation.
* Essential Thrombocythemia (all 6 criteria required)

  1. Platelets count ≥ 450 x 10 to 9/L
  2. Megakaryocyte proliferation with large and mature morphology. No significant increase or left shift of neutrophil granulopoiesis or erythropoiesis. Patients may have up to and including 2+ marrow reticulin fibrosis (0, 1 or 2 on scale 0 -4).
  3. Not meeting WHO criteria for CML, PV, MDS, PMF or other myeloid neoplasm
  4. Demonstration of clonal cytogenetic marker or no evidence of reactive thrombocytosis.
  5. Absence of a leukoerythroblastic blood picture.
  6. May participate in study without presence of JAK2V617F.

     Patients must have high risk disease as defined below:

     High risk PV ANY ONE of the following:
     * Age ≥ 60 years
     * Previous documented thrombosis, erythromelalgia or migraine (severe, recurrent, requiring medications, and felt to be secondary to the MPN) either after diagnosis or within 10 years before diagnosis and considered to be disease related
     * Significant splenomegaly (> 5cm below the left costal margin on palpitation) or symptomatic splenomegaly (splenic infarcts or requiring analgesia)
     * Platelets ≥ 1000 x 10 to 9/L
     * Diabetes or hypertension requiring pharmacological therapy for > 6 months

     High risk ET ANY ONE of the following:
     * Age ≥ 60 years
     * Platelet count ≥ 1500 x 10 to 9/L
     * Previous documented thrombosis, erythromelalgia or migraine headaches (severe, recurrent, requiring medications, and felt to be secondary to the MPN) either after diagnosis or within 10 years before diagnosis and considered to be disease related
     * Previous hemorrhage related to ET
     * Diabetes or hypertension requiring pharmacological therapy for > 6 months

     Other Inclusion criteria (Both Strata)
     * Diagnosed less than 5 years prior to entry on trial
     * Never treated with cytoreductive drugs except hydroxyurea for up to 3 months maximum (phlebotomy, aspirin allowed, anagrelide allowed)
     * Age: ≥ 18 years (no upper limit)
     * Ability and willingness to comply with all study requirements
     * Signed informed consent to participate in this study.
     * Willing to participate in associated correlative science biomarker study
     * Serum creatinine ≤ 1.5 x upper limit of normal
     * ST and ALT ≤ 2 x upper limit of normal
     * No known PNH (paroxysmal nocturnal hemoglobinuria) clone
     * No concurrent hormonal oral contraceptive use

     Exclusion Criteria:

     (ANY of the following, both strata)
     * Known to meet the criteria for primary myelofibrosis (as opposed to ET) by WHO 2008
     * Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
     * Any contraindications to pegylated interferon or hydroxyurea
     * Presence of any life-threatening co-morbidity
     * History of active substance or alcohol abuse within the last year
     * Subjects who are pregnant, lactating or of reproductive potential and not practicing an effective means of contraception
     * History of psychiatric disorder (e.g. depression) Subjects with a history of mild depression may be considered for entry into this study, provided that a pretreatment assessment of the subject's affective status supports that the subject is clinically stable based on the investigator's normal practice for such subject.
     * History of autoimmune disorder (e.g. hepatitis)
     * Hypersensitivity to interferon alfa
     * Hepatitis B or C infection (HBV), or untreated systemic infection
     * Known HIV disease
     * Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration) or clinically relevant ophthalmological disorder (e.g. due to diabetes mellitus or hypertension)
     * History or other evidence of decompensated liver disease
     * History or other evidence of chronic pulmonary disease associated with functional limitation
     * Thyroid dysfunction not adequately controlled
     * Neutrophil count <1.5 x 10 to 9/L
     * JAK2 exon 12 mutation: PV that lacks the JAK2V617F mutation but is characterized by the exon 12 mutation.
     * Meets criteria for post PV or post ET-MF
     * Subjects with any other medical condition, which in the opinion of the investigator would compromise the results of the study by deleterious effects of treatment.
     * Previous exposure to any formulation of pegylated interferon
     * History of major organ transplantation
     * History of uncontrolled severe seizure disorder
     * Inability to give informed written consent
     * Total bilirubin >1.5 x ULN (patients that have an isolated indirect bilirubin that causes total bilirubin to be elevated beyond 1.5 x ULN due to documented Gilbert's syndrome or hemolysis may be included). No detectable PNH (paroxysmal nocturnal hemoglobinuria) clone where tested

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-09; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hoffman, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Claire Harrison, MD, Study Chair — Guy's and St Thomas' NHS Foundation Trust; Ruben Mesa, MD, Study Chair — Mayo Clinic; Jean-Jacques Kiladjian, MD, Study Chair — Hopitaux de Paris; Mary Frances McMullin, MD, Study Chair — Belfast Health and Social Care Trust; John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (25):
- United States (16):
  - Mayo Clinic, Scottsdale, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - The Palo Alto Clinic, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Emory Hospital, Atlanta, Georgia
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Geisinger Cancer Center, Danville, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Hopitaux de Paris, Paris, France
- Italy (5):
  - Ospedale Riuniti de Bergamo, Bergamo
  - University Of Florence, Florence
  - Ospedale San Maartino Genova, Genova
  - San Matteo Hospital, Pavia
  - Universita Cattolica del Sacro Cuore, Rome
- United Kingdom (3):
  - Belfast City Hospital, Belfast, Northern Ireland
  - Heart of England NHS Foundation Trust, Birmingham
  - Guy's and St. Thomas' NHS Foundation Trust, London

REFERENCES:
- [Derived] Thanarajasingam G, Bhatnagar V, Noble BN, Chen TY, Fiero MH, Hoffman R, Jeffery M, Mazza GL, Mascarenhas J, Mesa R, Murugappan M, Ross J, Sidana S, Warsame R, Kluetz PG, Dueck AC. Longitudinal graphics of patient-reported physical function in patients treated for hematologic malignancies. BMC Med Res Methodol. 2025 Aug 7;25(1):189. doi: 10.1186/s12874-025-02617-y. PMID 40775758
- [Derived] Mascarenhas J, Kosiorek HE, Prchal JT, Rambaldi A, Berenzon D, Yacoub A, Harrison CN, McMullin MF, Vannucchi AM, Ewing J, O'Connell CL, Kiladjian JJ, Mead AJ, Winton EF, Leibowitz DS, De Stefano V, Arcasoy MO, Kessler CM, Catchatourian R, Rondelli D, Silver RT, Bacigalupo A, Nagler A, Kremyanskaya M, Levine MF, Arango Ossa JE, McGovern E, Sandy L, Salama ME, Najfeld V, Tripodi J, Farnoud N, Penson AV, Weinberg RS, Price L, Goldberg JD, Barbui T, Marchioli R, Tognoni G, Rampal RK, Mesa RA, Dueck AC, Hoffman R. A randomized phase 3 trial of interferon-alpha vs hydroxyurea in polycythemia vera and essential thrombocythemia. Blood. 2022 May 12;139(19):2931-2941. doi: 10.1182/blood.2021012743. PMID 35007321
- [Derived] Yacoub A, Mascarenhas J, Kosiorek H, Prchal JT, Berenzon D, Baer MR, Ritchie E, Silver RT, Kessler C, Winton E, Finazzi MC, Rambaldi A, Vannucchi AM, Leibowitz D, Rondelli D, Arcasoy MO, Catchatourian R, Vadakara J, Rosti V, Hexner E, Kremyanskaya M, Sandy L, Tripodi J, Najfeld V, Farnoud N, Papaemmanuil E, Salama M, Singer-Weinberg R, Rampal R, Goldberg JD, Barbui T, Mesa R, Dueck AC, Hoffman R. Pegylated interferon alfa-2a for polycythemia vera or essential thrombocythemia resistant or intolerant to hydroxyurea. Blood. 2019 Oct 31;134(18):1498-1509. doi: 10.1182/blood.2019000428. PMID 31515250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period from Sept 2011 through June 2016
Groups:
- PEGASYS: The subject received the PEGASYS at a dose level of 45 micrograms weekly and gradually increased to the maximum dose of 180 micrograms per week. The dose was administered by prefilled syringes and injected subcutaneously. Subjects received therapy for up to 12 months.
  Aspirin: Subject asked to take 81 to 100mg per day for the 12 months of the study treatment.
- Hydroxyurea: Subjects received a 500mg tablet to be taken twice daily for up to 12 months of treatment.
  Aspirin: Subject asked to take 81 to 100mg per day for the 12 months of the study treatment.
Period: Overall Study
Arm/Group | PEGASYS | Hydroxyurea
Started | 82 | 86
Completed | 13 | 12
Not Completed | 69 | 74
Not completed — Adverse Event | 12 | 9
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Treatment never started | 0 | 6
Not completed — Study closure by sponsor | 40 | 41
Not completed — Patient developed other disease | 0 | 1
Not completed — Transfer to another study | 0 | 1
Not completed — Unknown/missing | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEGASYS | Hydroxyurea | Total
Number analyzed (Participants) | 82 | 86 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (14.8) | 61.8 (12.8) | 59.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 49 | 49 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 4 | 7
  White | 76 | 70 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 8 | 11
Age > 60 years [Count of Participants; unit: Participants] | 42 | 56 | 98
The Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG measures level of functioning in terms of daily living abilities:
  0-Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg.light house work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about >50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair >50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 65 | 72 | 137
    1 | 15 | 13 | 28
    2 | 0 | 1 | 1
    3+ | 2 | 0 | 2
Disease Type [Count of Participants; unit: Participants]
  Essential thrombocythemia (ET) | 39 | 42 | 81
  Polycythemia Vera (PV) | 43 | 44 | 87
Previous Thrombosis [Count of Participants; unit: Participants] | 26 | 20 | 46
Previous Hemorrhage [Count of Participants; unit: Participants] | 3 | 4 | 7
Splenomegaly [Count of Participants; unit: Participants] | 5 | 6 | 11
Disease Duration [Median (Full Range); unit: months] | 2.6 [0 to 41.7] | 3.0 [0 to 84.2] | 2.8 [0 to 84.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission (CR)
Description: Number of participants with Complete Remission after 12 months of therapy assessed by hematologic response rates two strata of patients with high risk polycythemia vera (PV) or high risk essential thrombocythemia (ET). Complete remission means no evidence of disease.
Time Frame: 12 months
Population: there were 82 participants in PEGASYS arm 39 with ET and 43 with PV, 86 in Hydroxyurea arm 42 with ET and 44 with PV
Measure: Count of Participants; unit: Participants
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 82 | 86
Participants
  Essential Thrombocythemia: number analyzed (Participants) | 39 | 42
  Essential Thrombocythemia | 17 | 19
  Polycythemia Vera: number analyzed (Participants) | 43 | 44
  Polycythemia Vera | 12 | 13

2. Primary Outcome: Number of Participants With Partial Remission (PR)
Description: Number of participants with Partial Remission after 12 months of therapy assessed by hematologic response rates two strata of patients with high risk polycythemia vera (PV) or high risk essential thrombocythemia (ET). Partial Remission means decrease in the size of a tumor, or in the extent of cancer in the body, in response to treatment.
Time Frame: 12 months
Population: there were 82 participants in PEGASYS arm 39 with ET and 43 with PV, 86 in Hydroxyurea arm 42 with ET and 44 with PV
Measure: Count of Participants; unit: Participants
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 82 | 86
Participants
  Essential Thrombocythemia: number analyzed (Participants) | 39 | 42
  Essential Thrombocythemia | 10 | 11
  Polycythemia Vera: number analyzed (Participants) | 43 | 44
  Polycythemia Vera | 25 | 17

3. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 Hematological and Non-hematological Events
Description: Number of Participants with Grade 3 and Grade 4 Hematological and Non-hematological Events using the Common Terminology Criteria for Adverse Events (CTCAE) 4.0 to assess the toxicity, safety and tolerability of therapy (Pegylated Interferon Alfa-2a vs. Hydroxyurea).
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 82 | 86
Participants
  Grade 3 Hematological event | 3 | 2
  Grade 4 Hematological event | 0 | 0
  Grade 3 Non-hematological event | 27 | 14
  Grade 4 Non-hematological event | 2 | 3

4. Secondary Outcome: Change in the Total Symptom Score (TSS)
Description: Change in the Total Symptom Score which assessed improvement in disease symptoms measured by the change in TSS from the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) instrument being used in this study from baseline to 12 months. This 19 item instrument includes the previously validated 9 item brief fatigue inventory (BFI), symptoms related to splenomegaly, inactivity, cough, night sweats, pruritus, bone pains, fevers, weight loss, and an overall quality of life assessment. Each item is scored from 0-10 with full scale from 0-190, with higher scores mean worse symptoms.
Time Frame: baseline and 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 82 | 86
score on a scale | 1.16 [-2.04 to 4.36] | -1.0 [-4.38 to 2.39]

5. Secondary Outcome: JAK2 Allele Burden
Description: To compare the impact of therapy (Pegylated Interferon Alfa-2a vs. Hydroxyurea) on key biomarkers of the disease(s) by measuring the JAK2 allele burden.
Time Frame: 4 years
Population: data not collected
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Allele Burden
Description: The impact of PEGASYS on JAK2 will be measured by the allele burden; hematopoietic cell clonality will be measured by whether patients with clonal disease return to polyclonal; bone marrow histopathology will be measured by going from abnormal to normal; cytogenetic abnormalities will be measured by seeing if the cytogenetics go from abnormal to normal.To compare the impact of therapy on JAK2-V617F (JAK2), CALR, hematopoietic cell clonality in platelets and granulocytes in females, bone marrow histopathology, and cytogenetic abnormalities.
Time Frame: 4 years
Population: data not collected
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Progression of Disease or Death
Description: Survival and incidence of development of myelodysplastic syndrome, myelofibrosis, or leukemic transformation after therapy
  To estimate survival and incidence of development of myelodysplastic syndrome, myelofibrosis, or leukemic transformation after therapy (Pegylated Interferon Alfa-2a vs. Hydroxyurea) by capturing the rate of progression to a more advanced myeloid malignancy.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 82 | 86
Participants
  Death | 0 | 1
  Progression to MF | 0 | 0

8. Secondary Outcome: Number of Participants With Major Cardiovascular Events After Therapy
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | PEGASYS | Hydroxyurea
Number analyzed (Participants) | 82 | 86
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | PEGASYS | Hydroxyurea
All-Cause Mortality (participants affected / at risk) | 0/82 | 1/86
Serious Adverse Events (participants affected / at risk) | 14/82 | 4/86
Other Adverse Events (participants affected / at risk) | 79/82 | 76/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGASYS (N=82) | Hydroxyurea (N=86)
Bile Duct Disorder (Hepatobiliary disorders) | 1 | 0
Cardiac arrhythmias (Cardiac disorders) | 1 | 0
Cardiac disorder signs and symptoms (Cardiac disorders) | 1 | 0
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 1 | 0
Exocrine pancreas conditions (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrahges NEC (Gastrointestinal disorders) | 1 | 0
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 1 | 0
General system disorders NEC (General disorders) | 1 | 1
Headaches (Nervous system disorders) | 1 | 0
Infections - pathogen unspecified (Infections and infestations) | 0 | 2
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Platelet disorders (Blood and lymphatic system disorders) | 1 | 0
Pregnancy, labour, delivery and postpartum conditions (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Respiratory and mediastinal neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin and subcutaneous tissue infections and infestations (Skin and subcutaneous tissue disorders) | 1 | 0
Gallbladder disorders (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGASYS (N=82) | Hydroxyurea (N=86)
Abdominal Distenstion (Gastrointestinal disorders) | 0 | 1
Abdominal hernias and other abdominal wall conditions (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Administration site reactions (General disorders) | 15 | 0
Administration site reactions (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferace increased (Investigations) | 1 | 0
Allergic conditions (Immune system disorders) | 1 | 2
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 10 | 10
Anxiety (Psychiatric disorders) | 1 | 0
Anxeity disorders and symptoms (Psychiatric disorders) | 4 | 1
Appetite and general nutrition disorders (Metabolism and nutrition disorders) | 7 | 4
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Vascular disorders) | 1 | 2
Aural disorders NEC (Ear and labyrinth disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Back pain due to retroperitoneal fibrosis
Bacterial infectious disorders (Infections and infestations) | 7 | 4
Benign neoplasms gastrointestinal (Gastrointestinal disorders) | 0 | 1
Bladder and bladder neck disorders (excl calculi) (Renal and urinary disorders) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Body temperature conditions (General disorders) | 4 | 5
Bone and joint injuries (Injury, poisoning and procedural complications) | 6 | 0
Bone disorders (excl congenital and fractures) (Musculoskeletal and connective tissue disorders) | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone, calcium, magnesium and phosphorus metabolism disorders (Metabolism and nutrition disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Cardiac Signs and Symptoms NEC (Cardiac disorders) | 0 | 1
Cardiac and vascular investigations (excl enzyme tests) (Investigations) | 0 | 3
Cardiac arrhythmias (Cardiac disorders) | 1 | 3
Cardiac disorder signs and symptoms (Cardiac disorders) | 11 | 6
Central nervous system vascular disorders (Nervous system disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0 — Gastrointestinal nonspecific symptoms and therapeutic procedures (SMQ) Cardiomyopathy
Coagulopathies and bleeding diatheses (excl thrombocytopenic) (Blood and lymphatic system disorders) | 0 | 1
Cognitive and attention disorders and disturbances (Psychiatric disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Coronary artery disorders (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cranial nerve disorders (excl neoplasms) (Nervous system disorders) | 1 | 1
Cutaneous neoplasms benign (Skin and subcutaneous tissue disorders) | 1 | 0
Decreased and nonspecific blood pressure disorders and shock (Vascular disorders) | 2 | 3
Dental and gingival conditions (Gastrointestinal disorders) | 4 | 5
Depressed mood disorders and disturbances (Psychiatric disorders) | 11 | 1
Depression (Psychiatric disorders) | 1 | 2
Dermatitis and eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatology/skin, other (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Diarrhoea (excl infective) (Gastrointestinal disorders) | 0 | 1 — Gastrointestinal motility and defaecation conditions
Diverticular disorders (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 — Taste and smell disorders
Dysgeusia (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 4 | 4
Elevated ALT (Investigations) | 1 | 0
Endocrine disorders of gonadal function (Endocrine disorders) | 1 | 1
Enzyme investigations NEC (Investigations) | 2 | 0
Epidermal and Dermal Conditions (Skin and subcutaneous tissue disorders) | 0 | 1
Epidermal and Dermal Conditions (Skin and subcutaneous tissue disorders) | 24 | 19
Exocrine pancreas conditions (Gastrointestinal disorders) | 1 | 0
Eye disorders NEC (Eye disorders) | 6 | 3
Fatigue (General disorders) | 3 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 0
Fatigue or Tiredness (General disorders) | 0 | 1
Fatigue or Tiredness (General disorders) | 0 | 2
Flu-like symptoms (General disorders) | 0 | 1
Fungal infectious disorders (Infections and infestations) | 1 | 0
Gallbladder disorders (Hepatobiliary disorders) | 1 | 0
Gastrointestinal conditions NEC (Gastrointestinal disorders) | 1 | 0
Gastrointestinal infections (Gastrointestinal disorders) | 0 | 3
Gastrointestinal inflammatory conditions (Gastrointestinal disorders) | 1 | 1
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 16 | 20
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 24 | 18
Gastrointestinal stenosis and obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal vascular conditions (Gastrointestinal disorders) | 0 | 1
General malaise (General disorders) | 1 | 0
General system disorders NEC (General disorders) | 50 | 42
Genitourinary tract disorders NEC (Renal and urinary disorders) | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Glucose metabolism disorders (incl diabetes mellitus) (Endocrine disorders) | 4 | 3
Glucose metabolism disorders (incl diabetes mellitus) (Metabolism and nutrition disorders) | 4 | 2
Haematology investigations (incl blood groups) (Investigations) | 11 | 12
Haematopoietic neoplasms (excl leukaemias and lymphomas) (Blood and lymphatic system disorders) | 0 | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 11
Hearing disorders (Ear and labyrinth disorders) | 0 | 1
Heart failures (Cardiac disorders) | 1 | 1
Hepatic and hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 0 | 1
Hepatobiliary investigations (Investigations) | 12 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Infections - Pathogen Unspecified (Infections and infestations) | 0 | 1
Infections - pathogen class unspecified (Infections and infestations) | 0 | 1
Infections - pathogen unspecified (Infections and infestations) | 12 | 7
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 | 0
Injuries NEC (Injury, poisoning and procedural complications) | 3 | 4
Inner ear and VIIIth cranial nerve disorders (Ear and labyrinth disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Investigations, imaging and histopathology procedures NEC (Investigations) | 1 | 0
Joint Disorders (Musculoskeletal and connective tissue disorders) | 16 | 9
Lipid analyses (Investigations) | 3 | 1
Lipid metabolism disorders (Metabolism and nutrition disorders) | 4 | 2
Lymphocyte count decreased (Investigations) | 0 | 1
Lymphomas non-Hodgkin's T-cell (Blood and lymphatic system disorders) | 1 | 0
Male reproductive tract infections and inflammations (Reproductive system and breast disorders) | 2 | 0
Menstrual cycle and uterine bleeding disorders (Reproductive system and breast disorders) | 0 | 1
Mental impairment disorders (Nervous system disorders) | 1 | 2
Metabolic, nutritional and blood gas investigations (Investigations) | 2 | 3
Metabolic/laboratory, other (Metabolism and nutrition disorders) | 1 | 0
Middle ear disorders (excl congenital) (Ear and labyrinth disorders) | 0 | 3
Migraine (Nervous system disorders) | 1 | 0
Mood disorders and disturbances NEC (Psychiatric disorders) | 3 | 0
Movement disorders (incl parkinsonism) (Nervous system disorders) | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 0 | 2
Muscle disorders (Musculoskeletal and connective tissue disorders) | 9 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 — dystonia
Musculoskeletal and connective tissue deformities (incl intervertebral disc disorders) (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 17 | 17
Musculoskeletal and connective tissue neoplasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial disorders (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
nausea (Gastrointestinal disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — A disorder characterized by marked discomfort sensation in the neck area.
Malignant neoplasm of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous system disorders, unspecified (Nervous system disorders) | 0 | 1 — A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Neurological disorders NEC (Nervous system disorders) | 17 | 15
Neurological signs and symptoms NEC (Nervous system disorders) | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 0 — Blood/bone marrow
Non-cardiac chest pain (General disorders) | 1 | 1
Ocular haemorrhages and vascular disorders NEC (Eye disorders) | 2 | 0
Ocular infections, irritations and inflammations (Eye disorders) | 9 | 2
Ocular sensory symptoms NEC (Eye disorders) | 0 | 1
Ocular surface disease (Eye disorders) | 1 | 0
Oral soft tissue conditions (Gastrointestinal disorders) | 3 | 12
Skin disorders, Other (Skin and subcutaneous tissue disorders) | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Penile and scrotal disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 0 | 1
Peripheral neuropathies (Nervous system disorders) | 5 | 2
Physical examination topics (Investigations) | 1 | 1
Pigmentation disorders (Skin and subcutaneous tissue disorders) | 0 | 3
Platelet disorders (Blood and lymphatic system disorders) | 7 | 8
Procedural related injuries and complications NEC (Injury, poisoning and procedural complications) | 1 | 0
Prostatic disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 1 | 1
Protein and amino acid metabolism disorders NEC (Metabolism and nutrition disorders) | 1 | 0
Purine and pyrimidine metabolism disorders (Metabolism and nutrition disorders) | 4 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Renal and urinary tract investigations and urinalyses (Investigations) | 3 | 2
Renal and urinary tract neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal disorders (excl nephropathies) (Renal and urinary disorders) | 0 | 1
Reproductive neoplasms female benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 20 | 12
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Retina, choroid, and vitreous haemorrhages and vascular disorders (Eye disorders) | 0 | 1
Salivary gland conditions (Gastrointestinal disorders) | 5 | 2
Sensory Abnormalities NEC (Nervous system disorders) | 1 | 0
Sexual dysfunctions, disturbances and gender identity disorders (Psychiatric disorders) | 2 | 1
Sexual function and fertility disorders (Reproductive system and breast disorders) | 1 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders NEC (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue infections and infestations (Skin and subcutaneous tissue disorders) | 0 | 2
Skin appendage conditions (Skin and subcutaneous tissue disorders) | 8 | 7
Skin investigations (Investigations) | 0 | 1
Skin neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin vascular abnormalities (Skin and subcutaneous tissue disorders) | 2 | 2
Sleep disorders and disturbances (Psychiatric disorders) | 0 | 1
Sleep disturbances (incl subtypes) (Nervous system disorders) | 6 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 — Arthritis
Spleen, lymphatic and reticuloendothelial system disorders (Blood and lymphatic system disorders) | 2 | 0
Synovial and bursal disorders (Musculoskeletal and connective tissue disorders) | 2 | 2
Tendon, ligament and cartilage disorders (Musculoskeletal and connective tissue disorders) | 2 | 0
Thyroid gland disorders (Endocrine disorders) | 4 | 2
Tongue conditions (Gastrointestinal disorders) | 3 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Upper respiratory tract disorders (excl infections) (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Upper respiratory tract infections - pathogen class unspecified (Infections and infestations) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (Investigations) | 0 | 1
Urinary tract signs and symptoms (Renal and urinary disorders) | 3 | 3
Urolithiases (Renal and urinary disorders) | 1 | 0
Vascular disorders NEC (Vascular disorders) | 3 | 0
Vascular haemorrhagic disorders (Vascular disorders) | 1 | 3
Vascular hypertensive disorders (Vascular disorders) | 7 | 3
Venous varices (Vascular disorders) | 0 | 1
Viral infectious disorders (Infections and infestations) | 3 | 2
Vision disorders (Eye disorders) | 8 | 1
Vision disorders (Eye disorders) | 8 | 3
Vitamin related disorders (Metabolism and nutrition disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Water, electrolyte and mineral investigations (Investigations) | 2 | 0
White blood cell disorders (Blood and lymphatic system disorders) | 15 | 6
blurred vision (Eye disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
flu like symptoms (General disorders) | 1 | 0
headache (Nervous system disorders) | 1 | 0
kidney stone (Renal and urinary disorders) | 0 | 1
muscle, tendon, and ligament injuries (Injury, poisoning and procedural complications) | 0 | 1
rashes, eruptions, and exanthems NEC (Skin and subcutaneous tissue disorders) | 0 | 1
skin and subcutaneous conditions NEC (Skin and subcutaneous tissue disorders) | 0 | 1
skin appendage conditions (Skin and subcutaneous tissue disorders) | 0 | 1
skin appendage disorders (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT01259856/Prot_SAP_000.pdf